CLINICAL TRIAL: NCT03603418
Title: Role Of Dexamethasone In Induction Of Labor : A Randomized Clinical Trial .
Brief Title: Role Of Dexamethasone In Induction Of Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Kareem Medhat Mohamed Abdallah, ObGyn Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 292017
Record Dates: First submitted 2018-07-08; First posted 2018-07-27 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Dexamethasone Effect on Induction of Labor
MeSH Terms: interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Study group-Dexamethasone group) (Experimental): Forty patients undergoing induction of labor will receive 8 mg (2ml) of the product dexamethasone sodium phosphate intramuscular one hour before the initiation of labor induction in the form of epidrone ampoules which is a dexamethasone product from Epico-Egypt, and labor induction will be performed according to the American College of Obstetricians and Gynecologists protocol, i.e, starting by 25 mcg of PGE1 vaginally, in the form of Vagiprost, every 3-6 hours according to patient response, Dexamethasone will be given one hour before the first dose of Vagiprost, when bishop score reaches 6 to 8, oxytocin will be added by 5 drops/minute of 500 cc saline + 5 units of oxytocin with the dose increasing by 5-10 drops / minute every 30 minute till optimal contractions are reached which are three uterine contractions in 10 minutes and each lasting for 40-50 seconds
  Interventions: Drug: Dexamethasone Sodium Phosphate
- Group C (Control group) (Placebo Comparator): Forty patients undergoing induction of labor will receive 2ml of distilled water intramuscular one hour before the initiation of labor induction, and labor induction will be performed by the same protocol as above.
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate — Dexamethasone is a synthetic glucocorticoid that is commonly used in human medical practice as potent anti-inflammatory, immunosuppressive and analgesic agent.
  Arms: Group D (Study group-Dexamethasone group)
Other: Distilled water — Distilled water
  Arms: Group C (Control group)

SUMMARY:
Research hypothesis :

In pregnant women undergoing induction of labor, intramuscular injection of dexamethasone may accelerate induction delivery interval.

Research question :

In pregnant women undergoing induction of labor, does intramuscular injection of dexamethasone accelerate induction delivery interval ?

This study aims to assess the effect of intramuscular administration of dexamethasone on the induction delivery interval in full term patients undergoing induction of labor.

DETAILED DESCRIPTION:
The use of corticosteroids is one of the methods put forward for the strengthening and speeding up the process of labor. After identification of glucocorticoid receptors in human amnion, the role of corticosteroids in starting the process of labor has been studied in numerous studies. Some of them discussed the relation between dexamethasone injection and labor induction but still there is insufficient data. So by the end of this study it may be possible to assess the effect of intramuscular dexamethasone injection on shortening the induction delivery interval.

* Type of Study: Randomized Clinical Double Blind Trial .
* Study Setting: The study will be conducted at Ain Shams Maternity Hospital.
* Study Population: Full term patients who attend to the labor ward in El Demerdash Maternity Hospital and scheduled for induction of labor.
* Sample Size: Sample size was calculated using PASS® version 15.0, setting the power (β) at 0.02 and the significance level (α) at 0.05. Data from previous reports (Kashanian et al., 2008) indicated that mean Induction-Active phase Interval in women receiving 8mg of dexamethasone before induction of labor and controls was 3.09±1.5 and 4.21±1.8 hours respectively. Calculation according to these values produced a minimal sample size of 70 patients to be randomized equally to both groups. Assuming a drop-out rate of 15%, a minimum drop-out inflated enrollment sample size of approximately 80 women will be needed.
* Ethical Considerations: The study will be approved from the Ethical Committee of the Department of Obstetrics and Gynecology, Faculty of Medicine, Ain Shams University. Informed written consent will be taken from all women before recruitment in the study, and after extensive explanation and clear discussion of risks and benefits.
* Study Procedures: A total of 80 women undergoing induction of labor will be included in this study after taking their consent for this clinical trial after full explanation of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Primipara.
2. Gestational age (39-41) weeks according to Naegele's rule and a first-trimester ultrasound evaluation.
3. Vertex presentation.
4. Singleton fetus.
5. Intact fetal membranes.
6. No contraindication for vaginal delivery.
7. Cervix with a poor Bishop score (4-6).
8. Reactive CTG.
9. Average amount of liquor.

Exclusion Criteria:

1. Indication for cesarean section e.g. CPD, Placenta previa, IUGR, Non vertex presentation and previous cesarean section.
2. Maternal medical disorders as diabetes mellitus and severe pre-eclampsia.
3. Active phase of labor (cervical dilatation of 4 cm plus 3 forceful contractions over a ten minute span).
4. Preterm labor and premature rupture of membranes.
5. Multiparous women.
6. Significant vaginal bleeding. Placenta previa, probable placental abruption.
7. Fetal macrosomia>4.5 kg estimated by u/s.
8. Multiple pregnancy.
9. Fetal Distress and Non-reactive CTG.
10. Oligohydramnios.
11. IUGR.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Induction delivery interval | It may vary from 4 to 6 hours up to 72 hours
  The time between beginning of the induction of labor till the end of the 2nd stage of labor

SECONDARY OUTCOMES:
Induction active phase interval | It may vary from 2 to 3 hours up to 48 hours
  The time between beginning of the induction of labor till the beginning of the 1st stage of labor

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided